CLINICAL TRIAL: NCT02674711
Title: The Effect of a Brief Pre-operative Pain Medication Educational Video on Post-operative Prescription Opioid Medication Use in Patients Undergoing Spine Surgery. A Randomized Controlled Trial
Brief Title: Study of Opioid Use After Lumbar and Cervical Spine Surgery
Acronym: SOULCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: Baylor University (Other)
Responsible Party: Principal Investigator, Dan Rhon, Director of Physical Therapy, Center for the Intrepid, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.2015.048d
Record Dates: First submitted 2016-02-02; First posted 2016-02-04 (Estimated); Results first posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2022-07

CONDITIONS: Low Back Pain; Opiate Addiction; Neck Pain
Keywords: patient education; low back pain; post-surgical pain; chronic opioid use; Neck Pain
MeSH Terms: conditions — Low Back Pain; Opioid-Related Disorders; Neck Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Video (Experimental): Evidence-based video: Best Advice for People Taking Opioid Medication
  Interventions: Behavioral: Educational Video
- Usual Care (No Intervention): Usual care education provided at time of pre-operative appointment.

INTERVENTIONS:
Behavioral: Educational Video — The content of the education focus on providing a historical perspective for opioid prescription from the time when the risk of dependence was highly underestimated. The video discusses the current evidence for the effect of opioid medications in non-cancer non-acute pain. It also discusses some of the dangers of long-term opioid usage. The video is 11 and ½ minutes long.
  Other Names: Best Advice for People Taking Opioid Medication
  Arms: Educational Video

SUMMARY:
The purpose of this project is to assess the impact of an educational video on the use of prescription opioid medication during a 6-month period following spine surgery. Subjects will be recruited from the pool of patients coming in for the pre-operative appointment prior to spine surgery. Patients that consent and enroll will be randomized to receive either a brief educational video at this appointment or usual care. Patients will be followed after surgery weekly for the first month, and then again at 6 months to determine their prescription opioid medication utilization patterns. Prescription data will also be pulled from electronic medical records.

DETAILED DESCRIPTION:
After consenting, meeting inclusion criteria, and enrollment, all participants will complete several standard self-report questionnaires related to medical history, social demographic, and psychosocial variables that are related to low back pain, and often used in clinics that manage patients with low back pain. They will then be randomized to either receive the education, or only usual care (which is the typical information the surgeon provides the patient verbally during the pre-operative appointment). All patients will receive the usual care education from their surgeon.

Education Group:

The educational video is a white board style patient-centric video. The content of the education focus on providing a historical perspective for opioid prescription from the time when the risk of dependence was highly underestimated. The video discusses the current evidence for the effect of opioid medications in non-cancer on-acute pain. It also discusses some of the dangers of long-term opioid usage.

All Subjects:

All subjects will receive the usual care education that is typically given by their surgeon. That will be left up to the discretion of each surgeon.

All patients will proceed with the surgical procedure as planned. Each week during the 1-month period after the surgery, patients will be contacted, and then again at 6 months to ask history of prescription opioid utilization.

ELIGIBILITY:
Inclusion Criteria:

1. Currently scheduled for a pre-operative appointment with an orthopaedic spine surgeon or neurosurgeon specifically for a lumbar surgery.
2. Surgery is taking place for a condition that has been ongoing for 6 months or longer (chronic)
3. Between the age of 18 - 65 years
4. Read and speak English well enough to understand the education, provide informed consent and follow study instructions

Exclusion Criteria:

a. Known aversion or allergy that would prevent the patient from taking any opioid based pain medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rhon, DPT, DSc, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data sharing must first go through a Data Sharing Agreement approved by the Defense Health Agency.
Supporting Information: Study Protocol
Time Frame: Available for 1 year
Access Criteria: US Defense Health Agency data sharing agreement application approved
URL: https://www.health.mil/Military-Health-Topics/Privacy-and-Civil-Liberties/Submit-a-Data-Sharing-Application

REFERENCES:
- [Background] Manchikanti L, Abdi S, Atluri S, Balog CC, Benyamin RM, Boswell MV, Brown KR, Bruel BM, Bryce DA, Burks PA, Burton AW, Calodney AK, Caraway DL, Cash KA, Christo PJ, Damron KS, Datta S, Deer TR, Diwan S, Eriator I, Falco FJ, Fellows B, Geffert S, Gharibo CG, Glaser SE, Grider JS, Hameed H, Hameed M, Hansen H, Harned ME, Hayek SM, Helm S 2nd, Hirsch JA, Janata JW, Kaye AD, Kaye AM, Kloth DS, Koyyalagunta D, Lee M, Malla Y, Manchikanti KN, McManus CD, Pampati V, Parr AT, Pasupuleti R, Patel VB, Sehgal N, Silverman SM, Singh V, Smith HS, Snook LT, Solanki DR, Tracy DH, Vallejo R, Wargo BW; American Society of Interventional Pain Physicians. American Society of Interventional Pain Physicians (ASIPP) guidelines for responsible opioid prescribing in chronic non-cancer pain: Part 2--guidance. Pain Physician. 2012 Jul;15(3 Suppl):S67-116. PMID 22786449
- [Background] Trescot AM, Boswell MV, Atluri SL, Hansen HC, Deer TR, Abdi S, Jasper JF, Singh V, Jordan AE, Johnson BW, Cicala RS, Dunbar EE, Helm S 2nd, Varley KG, Suchdev PK, Swicegood JR, Calodney AK, Ogoke BA, Minore WS, Manchikanti L. Opioid guidelines in the management of chronic non-cancer pain. Pain Physician. 2006 Jan;9(1):1-39. PMID 16700278
- [Background] Devin CJ, Lee DS, Armaghani SJ, Bible J, Shau DN, Martin PR, Ehrenfeld JM. Approach to pain management in chronic opioid users undergoing orthopaedic surgery. J Am Acad Orthop Surg. 2014 Oct;22(10):614-22. doi: 10.5435/JAAOS-22-10-614. PMID 25281256
- [Background] Walid MS, Hyer L, Ajjan M, Barth AC, Robinson JS Jr. Prevalence of opioid dependence in spine surgery patients and correlation with length of stay. J Opioid Manag. 2007 May-Jun;3(3):127-8, 130-2. doi: 10.5055/jom.2007.0050. PMID 18027538
- [Background] Martell BA, O'Connor PG, Kerns RD, Becker WC, Morales KH, Kosten TR, Fiellin DA. Systematic review: opioid treatment for chronic back pain: prevalence, efficacy, and association with addiction. Ann Intern Med. 2007 Jan 16;146(2):116-27. doi: 10.7326/0003-4819-146-2-200701160-00006. PMID 17227935
- [Background] Deshpande A, Furlan A, Mailis-Gagnon A, Atlas S, Turk D. Opioids for chronic low-back pain. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD004959. doi: 10.1002/14651858.CD004959.pub3. PMID 17636781
- [Background] Lee D, Armaghani S, Archer KR, Bible J, Shau D, Kay H, Zhang C, McGirt MJ, Devin C. Preoperative Opioid Use as a Predictor of Adverse Postoperative Self-Reported Outcomes in Patients Undergoing Spine Surgery. J Bone Joint Surg Am. 2014 Jun 4;96(11):e89. doi: 10.2106/JBJS.M.00865. Epub 2014 Jun 4. PMID 24897746
- [Background] Chou R, Ballantyne JC, Fanciullo GJ, Fine PG, Miaskowski C. Research gaps on use of opioids for chronic noncancer pain: findings from a review of the evidence for an American Pain Society and American Academy of Pain Medicine clinical practice guideline. J Pain. 2009 Feb;10(2):147-59. doi: 10.1016/j.jpain.2008.10.007. PMID 19187891
- [Result] Rhon DI, Greenlee TA, Mayhew R, Boyer C, Laugesen M, Roth J, Dowd TC, Gill NW. Engaging Education About Risks of Opioid Use With Patients Before Elective Surgery of the Lower Extremity Did Not Reduce Postoperative Opioid Utilization: A Randomized Controlled Trial. J Am Acad Orthop Surg. 2022 Apr 1;30(7):e649-e657. doi: 10.5435/JAAOS-D-21-00603. PMID 35130200

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Educational Video | Usual Care
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Educational Video | Usual Care | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (11.0) | 45.5 (10.4) | 46.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 16 | 40
  Male | 36 | 44 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Other: American Indian or Alaska Native | 2 | 0 | 2
  Other: Asian | 2 | 1 | 3
  Other: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other: Black or African American | 14 | 12 | 26
  Other: White | 30 | 34 | 64
  Other: More than one race | 4 | 8 | 12
  Other: Unknown or Not Reported | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Opioid Medication Prescriptions
Description: Number of prescriptions within 12 months after surgery
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: prescriptions count
Arm/Group | Educational Video | Usual Care
Number analyzed (Participants) | 60 | 60
prescriptions count | 5.0 [3.8 to 6.7] | 5.1 [3.7 to 7.1]

2. Secondary Outcome: Modified Oswestry Disability Index (ODI) or Neck Disability Index (NDI)
Description: The ODI and NDI are 10-item scales with higher numbers indicating greater disability. Each item has 6 possible questions (0-5), which are then summed and multiplied to provide a % score out of 100%. The ODI focused on low back pain and the NDI on neck pain. As values are on the same scale, they were entered as one outcome since we included both neck and low back pain patients. Patients undergoing cervical spine surgery filled out the NDI (Neck Disability Index) and patients undergoing lumbar spine surgery filled out the ODI (Oswestry Disability Index)
Time Frame: 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Educational Video | Usual Care
Number analyzed (Participants) | 60 | 60
score on a scale | 41.7 [36.6 to 42.6] | 37.8 [33.0 to 42.6]

3. Secondary Outcome: Numeric Pain Rating Scale (NPRS)
Description: A 0-10 numeric pain rating scale ('0' indicating no pain, and '10' worst imaginable pain) will be used to assess pain intensity.
Time Frame: 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Educational Video | Usual Care
Number analyzed (Participants) | 60 | 60
score on a scale | 5.7 [5.0 to 6.5] | 5.1 [4.4 to 5.8]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Educational Video | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Educational Video (N=60) | Usual Care (N=60)
death (General disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/11/NCT02674711/Prot_SAP_000.pdf